CLINICAL TRIAL: NCT05581004
Title: A Phase Ia/Ib, Open Label, Multicenter, Dose-escalation Study to Evaluate the Safety, Pharmacokinetics, and Activity of RO7502175 as a Single Agent and in Combination With Checkpoint Inhibitor in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Activity of RO7502175 as a Single Agent and in Combination With Checkpoint Inhibitor in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO43860; 2021-006708-34 (EudraCT Number)
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced or Metastatic Solid Tumors; NSCLC; HNSCC; Melanoma; TNBC; Esophageal Cancer; Gastric Cancer; Cervical Cancer; Colorectal Cancer; Urothelial Carcinoma; Clear Cell RCC; HCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Melanoma; Esophageal Neoplasms; Stomach Neoplasms; Uterine Cervical Neoplasms; Colorectal Neoplasms; Carcinoma, Transitional Cell; Carcinoma, Renal Cell | interventions — atezolizumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase Ia: Dose Escalation (Experimental): Participants in successive cohorts will receive escalating doses of RO7502175, as an intravenous (IV) infusion on Day 1 of each 21-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: RO7502175
- Phase Ia: Expansion (Experimental): Participants with select solid tumors will receive a recommended dose of RO7502175, determined in Phase Ia Dose Escalation phase as an IV infusion on Day 1 of each 21-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: RO7502175
- Phase Ib: Dose Escalation (Experimental): Participants in successive cohorts will receive escalating doses of RO7502175, as an IV infusion, in combination with a fixed dose of atezolizumab, as an IV infusion on Day 1 of each 21-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: RO7502175; Drug: Atezolizumab
- Phase Ib: Expansion (Experimental): Participants with select solid tumors will receive a recommended dose of RO7502175, determined in Phase Ib Dose Escalation phase, as an IV infusion, in combination with a fixed dose of atezolizumab or pembrolizumab, as an IV infusion on Day 1 of each 21-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: RO7502175; Drug: Atezolizumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: RO7502175 — RO7502175 will be administered as per the schedules specified in the respective arms.
Drug: Atezolizumab — Atezolizumab will be administered as per the schedules specified in the respective arms.
  Arms: Phase Ib: Dose Escalation; Phase Ib: Expansion
Drug: Pembrolizumab — Pembrolizumab will be administered as per the schedules specified in the respective arms.
  Arms: Phase Ib: Expansion

SUMMARY:
This is a first-in-human study to evaluate the safety, tolerability, pharmacokinetics (PK), and anti-tumor activity of RO7502175 when administered as a single agent and in combination with atezolizumab or pembrolizumab in adult participants with locally advanced or metastatic solid tumors, including non-small-cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC), melanoma, triple-negative breast cancer (TNBC), esophageal cancer, gastric cancer, cervical cancer, colorectal cancer (CRC), urothelial carcinoma (UC), clear cell renal cell carcinoma (RCC) and hepatocellular carcinoma (HCC). Participants will be enrolled in 2 stages: dose escalation and dose expansion.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Measurable disease according to Response Evaluation criteria in Solid Tumors (RECIST) Version 1.1
* Histologically confirmed locally advanced, recurrent, or metastatic incurable solid tumor malignancy
* Tumor Specimen availability

Exclusion Criteria:

* Pregnant or breastfeeding or intention of becoming pregnant during the study or within 4 months after the final dose of RO7501275, or 4 months after the final dose of pembrolizumab, or 5 months after the final dose of atezolizumab
* Any anti-cancer therapy, whether investigational or approved, including chemotherapy, hormonal therapy, or radiotherapy, within 3 weeks prior to initiation of study treatment
* Active hepatitis B or C or tuberculosis
* Positive test for human immunodeficiency virus (HIV) infection
* Acute or chronic active Epstein-Barr virus (EBV) infection at screening
* Administration of a live, attenuated vaccine (e.g., FluMist) within 4 weeks before first RO7502175 infusion
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* Active or history of autoimmune disease
* Prior allogeneic stem cell or organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Number of Participants with Dose Limiting Toxicities (DLTs) | From Day 1 to Day 21 of Cycle 1 (21 days from date of first dose of study treatment)
Phase Ib: Number of Participants with DLTs | From Day 1 to Day 21 of Cycle 1 (21 days from date of first dose of study treatment)
Phase Ia: Number of Participants with Treatment Emergent Adverse Events | Up to approximately 5 years
Phase Ib: Number of Participants with Treatment Emergent Adverse Events | Up to approximately 5 years

SECONDARY OUTCOMES:
Phase Ia and Phase Ib: Maximum Serum Concentration (Cmax) of RO7502175 | From Cycle 1 (each cycle is 21 days) Day1 and at multiple timepoints up to each follow-up visits (up to approximately 5 years)
Phase Ia and Phase Ib: Objective Response Rate (ORR) | From Cycle 1(each cycle is 21 days) Day 1, until disease progression, death, or end of study (up to approximately 5 years)
Phase Ia and Phase Ib: Duration of Response (DOR) | From Cycle 1 (each cycle is 21 days) Day 1, until disease progression, death, or end of study (up to approximately 5 years)
Phase Ia and Phase Ib: Progression Free Survival (PFS) | From Cycle 1 (each cycle is 21 days) Day 1, until disease progression, death, or end of study (up to approximately 5 years)
Phase Ia and Phase Ib: Percentage of Participants With Anti-Drug Antibody (ADA) to RO7502175 | From Cycle 1 (each cycle is 21 days) Day 1 and at multiple timepoints up to treatment discontinuation (up to approximately 5 years)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (11):
  - Stanford University, San Francisco, California
  - University Of Colorado, Aurora, Colorado
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University Medical Center, Division of Oncology, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The West Clinic - Memphis (Union Ave), Germantown, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
- Australia (3):
  - Kinghorn Cancer Centre, Darlinghurst, New South Wales
  - Monash Health Monash Medical Centre, Clayton, Victoria
  - Linear Clinical Research Ltd, Nedlands, Western Australia
- Belgium (3):
  - UZ Antwerpen, Edegem
  - CHU de Liège, Herstal
  - GasthuisZusters Antwerpen, Wilrijk
- Canada (4):
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sir Mortimer B Davis Jewish General Hospital, Montreal, Quebec
- Greece (3):
  - University General Hospital ''ATTIKON'' - General Hospital of West Attica H AGIA VARVARA, Chaïdári, Attica
  - Papageorgiou General Hospital of Thessaloniki, N. Efkapria-Pavlos Melas, Thessaloniki
  - Sotiria Thoracic Diseases Hospital of Athens, Athens
- Netherlands (2):
  - Het Nederlands Kanker Instituut Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center - PPDS, Seoul
  - Samsung Medical Center - PPDS, Seoul
  - Severance Hospital Yonsei University Health System - Clinical Trials Center Pharmacy, Seoul
- Spain (6):
  - ICO l?Hospitalet ? Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Instituto de Investigacion Oncologica Vall dHebron (VHIO) - EPON, Barcelona
  - START MADRID_Hospital Universiario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario de Valencia, Valencia
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset Solna, Stokholm, Solna
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No